CLINICAL TRIAL: NCT00092612
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate Efficacy, Safety, and Tolerability of Ezetimibe 10 mg or Placebo Co-administered With Existing Simvastatin 10 mg or 20 mg in Attaining Low-Density Lipoprotein Cholesterol Target Levels in Patients With Hypercholesterolemia and Coronary Heart Disease.
Brief Title: Co-administration Study in Patients With Elevated Cholesterol and Coronary Heart Disease (0653-802)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-802; 2004_040
Record Dates: First submitted 2004-09-23; First posted 2004-09-27 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Coronary Disease
Keywords: Elevated Cholesterol
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0653, ezetimibe
Drug: Comparator: ezetimibe, placebo

SUMMARY:
The purpose of this study is to investigate additional cholesterol lowering effects in patients with coronary heart disease by giving an investigational drug with a patient's current approved cholesterol lowering medication.

DETAILED DESCRIPTION:
The duration of treatment is 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with elevated cholesterol and coronary heart disease

Exclusion Criteria:

* Patients who have cholesterol levels within normal ranges as identified by the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2003-05; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reaching their target LDL-C goal of </= 2.60 mmol/L, after 6 weeks of treatment

SECONDARY OUTCOMES:
Safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Farnier M, Volpe M, Massaad R, Davies MJ, Allen C. Effect of co-administering ezetimibe with on-going simvastatin treatment on LDL-C goal attainment in hypercholesterolemic patients with coronary heart disease. Int J Cardiol. 2005 Jul 10;102(2):327-32. doi: 10.1016/j.ijcard.2005.01.022. PMID 15982505